CLINICAL TRIAL: NCT05066880
Title: Investigation of the Effects of Yoga and Aerobic Exercise Training on Physical and Mental Health in People With Epilepsy
Brief Title: Yoga and Aerobic Exercise in Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Burcin Aktar, Institute of Health Sciences, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5258-GOA
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2022-12

CONDITIONS: Epilepsy; Epilepsy; Seizure; Epilepsy Idiopathic
Keywords: epilepsy; yoga; aerobic; exercise
MeSH Terms: conditions — Epilepsy; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga (Experimental): Participants allocated to the yoga group will receive the yoga-based intervention through an internet-based video conference remotely in real-time. Each class will accommodate a maximum of 5 subjects. A qualified physiotherapist who was a certificated yoga instructor will teach in these classrooms. The 8-week exercise intervention consists of three times per week sessions of yoga.
  Interventions: Other: Exercise training
- Aerobic exercise (Experimental): Participants of the aerobic exercise group will be requested to perform unsupervised aerobic training in the home environment (e.g., at home, park, backyard, or in the local gym). The 8-week exercise intervention consists of three times per week sessions of aerobic exercise. Training will consist of a 10-min warm-up period, aerobic activity, and 5-min cool-down period.
  Interventions: Other: Exercise training
- Wait-list (No Intervention): Participants in the wait-list group will be advised to continue their habitual physical activity next to usual medical care. A yoga or aerobic exercise program of 8 weeks will be offered after the ending of the study period.

INTERVENTIONS:
Other: Exercise training — Exercise training for 8 weeks
  Arms: Aerobic exercise; Yoga

SUMMARY:
In recent years, there is growing interest in illustrating the health benefits of exercise among epilepsy. Although exercise is recommended for patients with epilepsy, there is uncertainty concerning the effects of yoga and aerobic exercise on multiple health outcomes in epilepsy. The aim of this trial is to examine the effects of yoga and aerobic exercise training on physical activity, health-related physical fitness, mental, emotional, and psychological health status, seizure frequency and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epilepsy diagnosed by a neurologist using the International League Against Epilepsy (ILAE) criteria,
* Having access to the internet at least three per week.

Exclusion Criteria:

* Any history of neurological disorders other than epilepsy,
* Significant physical and cognitive impairments,
* Musculoskeletal comorbid conditions,
* Contraindications for an exercise intervention including diagnosed cardiovascular, pulmonary, or endocrine diseases,
* Pregnancy,
* Mental deficiency or low education level to understand the questionnaires,
* Currently participating in an exercise program,
* Volunteers who miss 3 consecutive intervention sessions, and do not participate in 10% of sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Physical activity in daily life | change from baseline to 8 weeks
  Physical activity will be objectively monitored with an accelerometer.
Seizure | change from baseline to 8 weeks
  Participants will be given a seizure diary and requested to record the number of their seizure.

SECONDARY OUTCOMES:
Six-Minute Walk test | change from baseline to 8 weeks
  The Six-Minute Walk test will be used to determine functional capacity.
30-second Chair Stand test | change from baseline to 8 weeks
  Lower body strength will be determined using the 30-second Chair Stand test.
Biodex Balance System | change from baseline to 8 weeks
  Balance evaluation will be performed with Biodex Balance System.
Bioelectrical impedance analyzer | change from baseline to 8 weeks
  Body composition measurements will be performed with bioelectrical impedance analyzer.
Waist and hip circumference | change from baseline to 8 weeks
  For the anthropometric measurements, waist and hip circumference will be taken.
Trail Making test and Digit Span test | change from baseline to 8 weeks
  The Trail Making test and Digit Span test will be used to evaluate for attention.
Stroop test and Verbal Fluency | change from baseline to 8 weeks
  The Stroop test and Verbal Fluency will be used to evaluate for executive functions.
Weschler Memory Scale-Revised Visual Reproduction subtest | change from baseline to 8 weeks
  The Weschler Memory Scale-Revised Visual Reproduction subtest will be used to evaluate for visual memory.
Clock Drawing test | change from baseline to 8 weeks
  The Clock Drawing test will be used to evaluate for visual perception and visual-spatial functions.
Oktem Verbal Memory Processes test | change from baseline to 8 weeks
  The Oktem Verbal Memory Processes test will be used to evaluate for verbal memory performance.
Neurological Disorders Depression Inventory for Epilepsy | change from baseline to 8 weeks
  The Neurological Disorders Depression Inventory for Epilepsy will be used to evaluate for depression.
Generalized Anxiety Disorder-7 | change from baseline to 8 weeks
  Anxiety will be determined by the Generalized Anxiety Disorder-7.
10-item Perceived Stress Scale | change from baseline to 8 weeks
  The 10-item Perceived Stress Scale will be used to assess subjective stress.
Fatigue Impact Scale | change from baseline to 8 weeks
  Fatigue will be assessed with the Fatigue Impact Scale.
Pittsburg Sleep Quality Index | change from baseline to 8 weeks
  Sleep quality will be measured using the Pittsburg Sleep Quality Index.
Quality of Life in Epilepsy Inventory-31 | change from baseline to 8 weeks
  It will be used to determine health-related quality of life for epilepsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aktar B, Balci B, Eraslan Boz H, Oztura I, Baklan B. Yoga and aerobic exercise in epilepsy: Study protocol for a randomized controlled trial. Physiother Res Int. 2023 Oct;28(4):e2013. doi: 10.1002/pri.2013. Epub 2023 May 7. PMID 37151132